CLINICAL TRIAL: NCT07019766
Title: National Longitudinal Cohort of Hematological Diseases-Large Granular Lymphocytic Leukemia
Acronym: NICHE-LGLL
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2025043
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: T-LGL Leukemia; NK-LGL Leukemia
Keywords: Treatment patterns; Hematologic response
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NICHE-LGLL: Patients who were diagnosed with LGLL in the investigating hospitals from Jan 1, 2000.
  Interventions: Other: A combined retrospective and prospective observational follow-up

INTERVENTIONS:
Other: A combined retrospective and prospective observational follow-up — The NICHE-LGLL will collect basic information, diagnostic and treatment information, as well as health costs information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

SUMMARY:
Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

The objectives of this study are to investigate the incidence and risk factors of large granular lymphocytic leukemia (LGLL) and to analyze the treatment effectiveness, patient prognosis, and healthcare costs in China.

1. Analyze the demographic and clinical characteristics of patients with LGLL, including sex, age, disease severity, and other relevant factors.
2. Examine disease features of LGLL patients, such as biochemical and hematological indicators, LGL counts, clonality, bone marrow pathology, and cytogenetics
3. Assess treatment patterns and real-world effectiveness in LGLL patients.
4. Evaluate clinical outcomes, including hematologic response, relapse, and mortality
5. Investigate long-term prognosis, including post-discontinuation outcomes and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with LGLL.
* Subjects treated at the Institute of Hematology and Blood Diseases Hospital from Jan 1, 2000.

Exclusion Criteria:

* Subject unlikely to be available for long-term follow-up for any reason (e.g., inability to obtain follow-up data or presence of severe comorbidities).
* Subject with alcohol or drug dependence that may reduce their compliance with the study.
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pantients diagnosed as LGLL.
  Diagnostic criteria for LGLL (Large Granular Lymphocytic Leukemia):
  Increased number of circulating LGL cells (>0.5×10^9/L) identified based on complete blood count and/or a consistent immunophenotypic pattern; Evidence of clonality confirmed by flow cytometry and/or molecular biology techniques; In patients with a low LGL cell count, diagnosis can still be made if there is a characteristic immunophenotype, STAT3 mutation, or bone marrow pathology abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2070-12-31 (Estimated); Study Completion 2070-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematologic response | Assessments will be conducted at baseline, 6 months, 12 months, and 24 months after treatment, as well as at study completion, with an average interval of approximately 1 year.
  Hematologic response contains improvements in neutrophil count, hemoglobin level, and platelet count

CONTACTS AND LOCATIONS:
Locations (1):
- Red Blood Cell Diseases Center and Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No